CLINICAL TRIAL: NCT03313427
Title: Early Physical Therapy Intervention in Preterm Infants During the Stay in the Neonatal Intensive Care Unit and at Home to Promote Motor Development
Brief Title: Early Physical Therapy Intervention in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vic - Central University of Catalonia (Other)
Collaborators: Hospital Sant Joan de Deu (Other)
Responsible Party: Principal Investigator, Mirari Ochandorena Acha, Physiotherapist, MSc, PhD St., University of Vic - Central University of Catalonia
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: PTNEO-001
Record Dates: First submitted 2017-10-09; First posted 2017-10-18 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Preterm Infant; Physical Therapy; Early Intervention; NICU; Home; Motor Development
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Usual care Early physical therapy intervention at the UCIN and after discharge, at home; based on the family-centered model.
  Interventions: Other: Physical Therapy Early Intervention
- Control (Other): Usual care
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Physical Therapy Early Intervention — At the UCIN:
  * Parental education to empower them on motor development and parent-infant relationship. Consisted on 6 sessions during the first weeks at the NICU.
  * Tactile and kinaesthetic stimulation managed by parents. 2 times a day, 15 minutes each, during 10 days.
  At home:
  Psychomotor Development Program for the baby; comprised of different exercises, in different phases, depending on child maturation stage. Started after hospital discharge until 2 months corrected age.
  Arms: Intervention
Other: Usual Care — NICU usual care
  Arms: Control

SUMMARY:
The hypothesis of this study is that early physical therapy intervention, initiated during the NICU stay and up to 2 months corrected age, based on the family-centered model, could promote preterm infants motor development in short-term (2 months corrected age) and long-term (8 months corrected age).

There is a high evidence level of different systematic reviews, which support the effectivity of early intervention with preterm infants.

The principal aim of this randomized controlled trial is to evaluate the effectiveness of early physiotherapy intervention to promote motor development in preterm infants at 2 and 8 months corrected age.

The secondary purpose is to study the motor development of those preterm infants who received early physical therapy intervention.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants, gestational age between 28-34 weeks
* Families with ability to take care of the child, without chronic or mental illness
* Long-term parental presence in the hospital (at least 10h/day)

Exclusion Criteria:

* Children diagnosed with congenital disease or brain injury (LPV, HIV), before or during the study
* Children undergoing major surgery (cardiac intervention, Ductus, thoracic intervention)
* Children with musculoskeletal deformities

Ages: 28 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Motor development. | 2 months corrected age and 8 months corrected age
  Assessed by the Alberta Infant Motor Scale (AIMS). Total maximum score 40 points. Higher values represent a better outcome.

SECONDARY OUTCOMES:
Movement quality. | 40 weeks postmenstrual age and 2 months corrected age
  Assessed by the General Movements Assessment. The assessment provide the quality of the movement (suboptimal/optimal/pathological).
Gross motor and fine motor function. | 8 months corrected age
  Assessed by the Bayley Scale of Infant Development III. Percentile ranks from 1 to 99. Higher percentile represent a better outcome
Development and risk of development delay. | 1 months corrected age and 8 months corrected age
  Assessed by the Ages and Stages Questionnaires Third Edition (ASQ-3). 30 questions covering 5 domains of development: communication, gross motor, fine motor, problem-solving and adaptive skills.
Mothers' stress index. | after the intervention, 3 months corrected age
  Assessed by the Parents Stress Index - Short Form. Composed of 36 items with a Likert-type answer format of five options.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Sant Joan de Deu, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ochandorena-Acha M, Terradas-Monllor M, Lopez Sala L, Cazorla Sanchez ME, Fornaguera Marti M, Munoz Perez I, Agut-Quijano T, Iriondo M, Casas-Baroy JC. Early Physiotherapy Intervention Program for Preterm Infants and Parents: A Randomized, Single-Blind Clinical Trial. Children (Basel). 2022 Jun 15;9(6):895. doi: 10.3390/children9060895. PMID 35740832